CLINICAL TRIAL: NCT03349723
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses of BI 1265162 in Healthy Male Volunteers in a Partially Randomised, Single Blind, Placebo-controlled Trial
Brief Title: This Study Tests the Safety, Tolerability and How Different Doses of BI 1265162 Are Taken up in the Body of Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1399-0001; 2017-001106-15 (EudraCT Number)
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1265162 (Experimental): BI 1265162
  Interventions: Drug: BI 1265162
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1265162 — Single rising dose groups
  Arms: BI 1265162
Drug: Placebo — Single rising dose groups
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1265162 in healthy male subjects following inhalative administration of single rising doses.

Secondary objective is the exploration of the pharmacokinetics (PK) of BI 1265162 after single dosing.

DETAILED DESCRIPTION:
To investigate safety, tolerability and pharmacokinetics of BI 1265162 in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Forced Expiratory Volume in one second (FEV1) and Forced Vital Capacity (FVC) of equal or greater than 80% of predicted normal, at screening and prior to randomisation
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* A history of chronic kidney disease (EGFR <59 mls/min including corrections as per ethnicity)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* The subject has a diagnosis history of pulmonary hyperreactivity
* Male subjects with woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 14 days after last administration of trial medication (BI 1265162 or placebo)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was single-blind, partially randomised, and placebo controlled within parallel dose groups trial. A total of 57 participants were entered and 56 were treated. The dose range for Treatment A to Treatment G was 3 μg to 1200 μg.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- 3 Microgram BI 1265162: 3 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 10 Microgram BI 1265162: 10 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 30 Microgram BI 1265162: 30 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 100 Microgram BI 1265162: 100 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 300 Microgram BI 1265162: 300 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 600 Microgram BI 1265162: 600 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- 1200 Microgram BI 1265162: 1200 microgram BI 1265162 solution for inhalation was administered orally via Respimat® inhaler.
- Placebo Matching BI 1265162: Subjects administered single dose of placebo matching BI 1265162 solution for inhalation orally via Respimat® inhaler.
Period: Overall Study
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162 | Placebo Matching BI 1265162
Started (Started are the Treated) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set(TS):This subject set included all subjects who had received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162 | Placebo Matching BI 1265162 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (3.6) | 31.8 (5.2) | 28.7 (4.7) | 44.7 (5.6) | 32.0 (7.3) | 34.5 (8.9) | 38.8 (9.8) | 35.1 (11.0) | 34.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 14 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs)
Description: Percentage of participants with drug-related adverse events (AEs).
Time Frame: From drug administration until end of trial examination, up to 9 days
Population: Treated set(TS): This subject set included all subjects who had received at least 1 dose of trial medication.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162 | Placebo Matching BI 1265162
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Percentage of participants (%) | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 0

2. Secondary Outcome: Maximum Measured Concentration of BI 1265162 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1265162 in plasma (Cmax).
Time Frame: Pharmacokinetic samples were taken pre-dose and 0:02 (hour: minute), 0:05, 0:10, 0:15, 0:20 , 0:30, 0:45, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 48:00 and 72:00 (Last time point only taken for 1200 µg) after drug administration
Population: The Pharmacokinetic set (PKS) included all subjects of the TS who received BI 1265162 and provided at least 1 PK parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles Per Litre (pmol/L)
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Picomoles Per Litre (pmol/L) | 17.8 (32.9) | 50.1 (46.6) | 129.0 (40.1) | 462.0 (53.2) | 1090.0 (26.0) | 3130.0 (30.6) | 6500.0 (73.1)
Statistical Analysis 1: Comparison: 3 Microgram BI 1265162 vs 10 Microgram BI 1265162 vs 30 Microgram BI 1265162 vs 100 Microgram BI 1265162 vs 300 Microgram BI 1265162 vs 600 Microgram BI 1265162 vs 1200 Microgram BI 1265162; The model consisted of a regression model applied to log-transformed data. The corresponding ANCOVA model included the logarithm of the dose as a covariate; Test type: Other; Slope = 0.9806, 95% CI 2-sided [0.9155 to 1.0457], Standard Error of Mean 0.0322 — Based on the estimate for the slope parameter (β), a 2-sided 95% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1

3. Secondary Outcome: Area Under the Concentration-time Curve of the BI 1265162 in Plasma Over the Time Interval 0 to 1 Hour Post-dose (AUC0-1)
Description: Area under the concentration-time curve of the BI 1265162 in plasma over the time interval 0 to 1 hour post-dose (AUC0-1)
Time Frame: Pharmacokinetic samples were taken pre-dose and 0:02 (hour: minute), 0:05, 0:10, 0:15, 0:20 , 0:30, 0:45, 1:00 after drug administration
Population: The Pharmacokinetic set (PKS) included all subjects of the TS who received BI 1265162 and provided at least 1 PK parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability. Only subjects with non-missing values were included in the analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles*Hour Per Litre (pmol*h/L)
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
Picomoles*Hour Per Litre (pmol*h/L) | 10.4 (42.4) | 28.7 (49.0) | 73.7 (43.4) | 299.0 (45.2) | 706.0 (25.9) | 1700.0 (34.5) | 3920.0 (76.4)
Statistical Analysis 1: Comparison: 3 Microgram BI 1265162 vs 10 Microgram BI 1265162 vs 30 Microgram BI 1265162 vs 100 Microgram BI 1265162 vs 300 Microgram BI 1265162 vs 600 Microgram BI 1265162 vs 1200 Microgram BI 1265162; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.9892, 95% CI 2-sided [0.9207 to 1.0577], Standard Error of Mean 0.0339 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From drug administration until end of trial examination, up to 9 days.
Arm/Group | 3 Microgram BI 1265162 | 10 Microgram BI 1265162 | 30 Microgram BI 1265162 | 100 Microgram BI 1265162 | 300 Microgram BI 1265162 | 600 Microgram BI 1265162 | 1200 Microgram BI 1265162 | Placebo Matching BI 1265162
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6 | 1/6 | 2/6 | 0/6 | 1/6 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 Microgram BI 1265162 (N=6) | 10 Microgram BI 1265162 (N=6) | 30 Microgram BI 1265162 (N=6) | 100 Microgram BI 1265162 (N=6) | 300 Microgram BI 1265162 (N=6) | 600 Microgram BI 1265162 (N=6) | 1200 Microgram BI 1265162 (N=6) | Placebo Matching BI 1265162 (N=14)
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03349723/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03349723/SAP_001.pdf